CLINICAL TRIAL: NCT07218172
Title: Characterization and Clinical Outcomes of Severe Asthma Patients in Israel Treated With Benralizumab (SAIL-B)
Acronym: SAIL-B
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00126
Record Dates: First submitted 2025-09-29; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective, observational, one arm, single country study, using the computerized database of Maccabi Health Services (MHS). The study will include adult patients who initiated benralizumab treatment for SEA between January 1, 2019, and March 31, 2024. The study population will include both biologic-naive and biologic-experienced patients. Patients will be followed from 12 months before the index date until the earliest of the following dates: switching, death, leaving MHS or end of the study follow-up period (June 30, 2024).

ELIGIBILITY:
Inclusion Criteria:

* An authorization from MHS drugs authorization center for benralizumab, with a diagnosis of asthma (ICD-9 code 493.X and the corresponding internal MHS diagnosis codes for SA). Having an authorization indicates that patients have severe eosinophilic asthma and fulfil the GINA definition of severe asthma as well as additional local reimbursement criteria.
* At least one purchase of benralizumab for the first time between January 1 2019 and March 31 2024.
* Age ≥18 years on the index date.
* MHS members for at least 12 months before the index date.

Exclusion Criteria:

• Patients who received benralizumab for indication other than asthma according to MHS drugs authorization center.

- currently or recently included in a clinical trial according to the ICD-9 diagnosis code V70.7) and the corresponding internal MHS codes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult patients who initiated benralizumab treatment for SEA between January 1, 2019, and March 31, 2024. The study population will include both biologic-naive and biologic-experienced patients
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Asthma related characteristics | Jan2019-Mar2024
  Number of exacerbations (baseline)

SECONDARY OUTCOMES:
Asthma related measure | Jan2019-Mar2024
  Number of asthma exacerbations during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Tel Aviv, Israel